CLINICAL TRIAL: NCT03241264
Title: A Phase 1, Open-Label, Randomized-Sequence, Single-Crossover, Bridging Study to Evaluate the Single-Dose Pharmacokinetics, Safety, and Tolerability of Two ND-L02-s0201 Formulations, Frozen Versus Lyophilized, Administered by Intravenous Infusion to Healthy Male and Female Subjects
Brief Title: A Study of Safety, Tolerability, and the Effects Two ND-L02-s0201 Have on the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nitto Denko Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ND-L02-s0201-004
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module A (Experimental): Lyophilized Formulation
  Interventions: Drug: ND-L02-s0201
- Module B (Experimental): Frozen Formulation
  Interventions: Drug: ND-L02-s0201

INTERVENTIONS:
Drug: ND-L02-s0201 — Specified dose on specified day

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and the effects two ND-L02-s0201 have on the body

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health, as determined by the Investigator
* Subject consumes an average of no more than 2 alcoholic drinks per day within the 6 months before administration of study drug
* Subject has serum calcium and parathyroid hormone (intact) within the limits of the normal range of the laboratory

Exclusion Criteria:

* Subject has a disease or condition (medical or surgical) which, in the opinion of the Investigator, may compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, or central nervous systems; or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of ND-L02-s0201 solution, or that may place the subject at increased risk
* Subject has a history of bone disease, including osteoporosis and osteomalacia, Paget's disease of bone, or a history of unexplained fractures or fractures after minimal trauma
* Subject has abnormal laboratory values considered to be clinically significant by the Investigator

Other protocol inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 28 days
Time to maximum plasma concentration (Tmax) | Up to 28 days
Area under the plasma concentration-time curve from time 0 to the last available observable concentration (AUC0-t) | Up to 28 days
Area under the plasma concentration-time curve extrapolated to infinity (AUC0-∞) | Up to 28 days
Area under the first moment of the plasma concentration-time curve from time zero to infinity (AUMC0-inf) | Up to 28 days
Apparent first-order terminal elimination rate constant (Kel) | Up to 28 days
Volume of distribution during the elimination phase after IV administration (Vz) | Up to 28 days
Apparent volume of distribution at steady-state (Vss) | Up to 28 days
Total plasma clearance of drug after IV administration (CL/F) | Up to 28 days
Apparent first-order terminal elimination half-life (T1/2) | Up to 28 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 28 days
Incidence of serious adverse events (SAEs) | Up to 28 days
Incidence of discontinuations of study drug due to toxicity | Up to 28 days